CLINICAL TRIAL: NCT05861284
Title: Developing and Optimizing Transcranial Magnetic Stimulation for Motor Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elisa Kallioniemi (Other)
Responsible Party: Sponsor-Investigator, Elisa Kallioniemi, Assistant Professor, New Jersey Institute of Technology
Organization: New Jersey Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB_2303032088
Record Dates: First submitted 2023-04-27; First posted 2023-05-16 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Motor Cortex; Motor Skills
Keywords: TMS; Motor system; Healthy
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single-pulse TMS over the primary motor cortex (Experimental): We will administer single-pulse TMS to the primary motor cortex while measuring motor responses and just before a skill-learning task.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Paired-pulse TMS over the primary motor cortex (Experimental): We will administer paired-pulse TMS to the primary motor cortex while measuring motor responses and just before a skill-learning task.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Sham TMS over the primary motor cortex (Sham Comparator): We will administer sham TMS to the primary motor cortex while measuring motor responses and before a skill-learning task.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Transcranial magnetic stimulation (TMS) is a non-invasive brain stimulation method that can induce long-term changes in connections between neuronal networks.

SUMMARY:
This study aims to evaluate three different transcranial magnetic stimulation protocols and their impact on motor system neurophysiology and skill learning.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) is a non-invasive brain stimulation method that induces long-term changes in connections between neuronal networks. This and the ability to activate the whole motor system allows the use of TMS to facilitate motor recovery. The motor system has different excitatory states associated with ongoing mu oscillation. Here, the investigators will monitor brain mu oscillations in real-time non-invasively using electroencephalography and modulate the function of the motor system. The investigators will test the impact of three different TMS protocols on motor system neurophysiology and skill learning. These data will provide novel understanding needed to improve TMS approaches for individuals requiring motor rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* Able to read, understand, and sign the informed consent in English
* Right-handed

Exclusion Criteria:

* A sensory or physical impairment
* History of epilepsy or seizures in the family
* Non-removable metal or electronics (e.g., a cochlear implant, cardiac pacemaker, or implanted electronic devices) in your head or body
* A head injury with loss of consciousness
* Diagnosis of psychiatric or neurological disorder
* Skin defects or active infections on the scalp or hands
* Pregnancy or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Effect of TMS on motor evoked potentials | Up to 1 second after TMS
  Amplitude of the motor evoked potentials in millivolts.
Skill learning accuracy | Up to 12 minutes
  Skill learning accuracy as the total number of correct responses.
Skill learning speed | Up to 12 minutes
  Skill learning speed in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Kallioniemi, Ph.D., Principal Investigator — New Jersey Institute of Technology

IPD SHARING:
Plan to Share IPD: Yes
Preprocessed and anonymized data will be provided upon request to the faculty / research staff of recognized research, medical, and educational institutions for educational and scientific purposes.
Supporting Information: Study Protocol
Time Frame: Data will be shared only upon request after the study has ended (within 6 months).
Access Criteria: To receive access, the study investigators must be contacted via an institutional e-mail.